CLINICAL TRIAL: NCT05632991
Title: Ultrasound Guided External Oblique Intercostal Plane Block vs. Transversus Abdominis Plane Block for Laparoscopic Cholecystectomy: Prospective Randomized Study
Brief Title: External Oblique Intercostal Plane Block vs. Transversus Abdominis Plane Block for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ataunilapcholecystectomy
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External oblique intercostal plane block (Active Comparator): Ultrasound-guided External oblique intercostal plane block before surgery
  Interventions: Other: ultrasound guided external oblique intercostal plane block
- Subcostal Transversus Abdominis Plan Block Group (Active Comparator): Ultrasound-guided Subcostal Transversus Abdominis Plan Block Group
  Interventions: Other: Subcostal Transversus Abdominis Plan Block Group

INTERVENTIONS:
Other: ultrasound guided external oblique intercostal plane block — ultrasound guided external oblique intercostal plane block 20 ml local anesthetic each side
  Arms: External oblique intercostal plane block
Other: Subcostal Transversus Abdominis Plan Block Group — ultrasound guided Subcostal Transversus Abdominis Plan Block Group 20 ml local anesthetic each side
  Arms: Subcostal Transversus Abdominis Plan Block Group

SUMMARY:
The laparoscopic approach has become the gold standard for many abdominal surgical procedures, including cholecystectomy. Compared to laparotomy, laparoscopy allows smaller incisions, reduces perioperative stress response, reduces postoperative pain, and results in shorter recovery time.

However, anaesthesia concerns in patients undergoing laparoscopic surgery are different from patients undergoing open abdominal surgery.

The aim of this study is to investigate the effect of the external oblique intercostal block, which is a new block, on postoperative pain score and opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients
* Laparoscopic cholecystectomy

Exclusion Criteria:

* Chronic pain bleeding disorders renal or hepatic insufficiency patients on chronic non-steroidal anti-inflammatory medications emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | first 24 hours
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | postextubation 0-24 hours
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Woldu SL, Weinberg AC, Bergman A, Shapiro EY, Korets R, Motamedinia P, Badani KK. Pain and analgesic use after robot-assisted radical prostatectomy. J Endourol. 2014 May;28(5):544-8. doi: 10.1089/end.2013.0783. Epub 2014 Jan 30. PMID 24400824
- [Background] Leitao MM Jr, Malhotra V, Briscoe G, Suidan R, Dholakiya P, Santos K, Jewell EL, Brown CL, Sonoda Y, Abu-Rustum NR, Barakat RR, Gardner GJ. Postoperative pain medication requirements in patients undergoing computer-assisted ("Robotic") and standard laparoscopic procedures for newly diagnosed endometrial cancer. Ann Surg Oncol. 2013 Oct;20(11):3561-7. doi: 10.1245/s10434-013-3064-9. PMID 23797751
- [Derived] Al S, Ahiskalioglu A, Karapinar YE, Yayik AM, Aydin ME, Celik EC, Ahiskalioglu EO, Doymus O. External oblique intercostal plane block as an alternative to subcostal TAP block for laparoscopic cholecystectomy: a prospective randomized study. BMC Anesthesiol. 2025 Dec 5;26(1):26. doi: 10.1186/s12871-025-03548-3. PMID 41351140